CLINICAL TRIAL: NCT00538902
Title: A Multi-center Randomized, Phase 2/3, Double-blind, Parallel-group, Placebo-controlled Study to Assess the Safety and Efficacy of Adalimumab Administered as Subcutaneous Injections in Adult Chinese Rheumatoid Arthritis Subjects Treated With Methotrexate
Brief Title: Safety and Efficacy Study of Adalimumab in Adult Chinese Rheumatoid Arthritis Subjects Treated With Methotrexate
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Laura Redden MD, PhD, Project Director, Abbott
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M04-705
Record Dates: First submitted 2007-10-01; First posted 2007-10-03 (Estimated); Results first posted 2009-12-30 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Humira, methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo administered subcutaneously every other week
  Interventions: Biological: Placebo
- Adalimumab 80 mg (Experimental): Adalimumab 80 mg administered subcutaneously every other week
  Interventions: Biological: Adalimumab 80 mg
- Adalimumab 40 mg (Experimental): Adalimumab 40 mg administered subcutaneously every other week
  Interventions: Biological: Adalimumab 40 mg

INTERVENTIONS:
Biological: Placebo — Placebo administered subcutaneously (SC) every other week (eow) for 12 weeks, followed by adalimumab 40 mg SC eow for 92 weeks.
  Arms: Placebo
Biological: Adalimumab 80 mg — Adalimumab 80 mg administered subcutaneously (SC) every other week (eow) for 12 weeks, followed by adalimumab 40 mg SC eow for 92 weeks.
  Other Names: Humira
  Arms: Adalimumab 80 mg
Biological: Adalimumab 40 mg — Adalimumab 40 mg administered subcutaneously every other week for 104 weeks
  Other Names: Humira
  Arms: Adalimumab 40 mg

SUMMARY:
A study to assess the safety and efficacy of adalimumab administered as a subcutaneous injection in adult Chinese subjects with rheumatoid arthritis and treated with methotrexate

DETAILED DESCRIPTION:
This was a multi-center, Phase 2/3, randomized, double-blind (DB), parallel group, placebo controlled, safety and efficacy study in adult Chinese RA subjects. The duration of the study was approximately 116 weeks. This included a 4-week (28 days) Screening period, a 12-week Double-Blind (DB) period, a 90-week Open-Label (OL) Period, and a 10-week (70 days) Follow-up period. The 70-day Safety Follow-up period was initiated after the last dose of study medication.

During the DB period, 302 Chinese subjects with RA and concomitantly treated with MTX were enrolled at 11 clinical sites located throughout China. Subjects were randomly assigned to one of the three treatment groups in a 2:2:1 ratio: 80 mg adalimumab, 40 mg adalimumab, or placebo. From Week 0 to Week 10, subjects received blinded study drug. Subjects who successfully participated and completed Week 12 of the DB portion of the study participated in the OL period. All subjects in the OL period received adalimumab 40 mg. Throughout the study, the study drug was administered subcutaneously (SC) every other week (eow).

Subjects that completed the Week 24 visit, prior to the approval of Protocol Amendment 1, had 70 days from the last dose of study drug to re-enter the study. The Investigator confirmed that the subject did not develop any of the exclusion criteria and completed the procedures defined by the OL Screening visit.

Results through Week 24 of this study were presented in the regulatory dossier for the marketing authorization application of Humira in China, fulfilling the requirement for clinical data in Chinese patients. However, in order to continue to provide treatment to patients who responded well to adalimumab, subjects had the option to continue in the OL extension of this study until Week 92.

ELIGIBILITY:
Inclusion Criteria:

* Met ACR criteria for diagnosis of active rheumatoid arthritis (RA) and have had at both the Screening visit and Week 0 visit at least four swollen joints (out of 66 assessed) and at least six tender joints(out of 68 assessed)
* Subjects must have failed prior treatment with one or more disease-modifying antirheumatic drugs (DMARDs)
* DMARDs (other than methotrexate [MTX]) must have been discontinued for >= 28 days or at least 5 half-lives, whichever is greater, before the Week 0 visit
* Traditional Chinese Medicines must have been discontinued for >= 28 days before the Week 0 visit
* Subjects must have received at least three months of treatment with MTX (minimum 7.5 mg/week) and remained on a stable dose of MTX for >= 28 days prior to the Screening visit
* Glucocorticoids equivalent to <= 10 mg of prednisone and prednisone equivalent must have remained unchanged for at least 28 days prior to the Week 0 visit
* Must have been able and willing to give written informed consent and to comply with the requirements of this study protocol

Exclusion Criteria:

* A history of, or current, acute inflammatory joint disease of different origin (e.g., mixed connective tissue disease, seronegative spondyloarthropathy, psoriatic arthritis, Reiter's syndrome, systemic lupus erythematosus, fibromyalgia or any arthritide with onset prior to age 16 years
* Wheelchair-bound or bedridden
* Joint surgery involving joints to be assessed within this study, within two months prior to the Screening visit
* Intra-articular, intramuscular or intravenous administration of corticosteroids within 28 days prior to the Screening visit
* Prior treatment with any TNF antagonist, including adalimumab
* Subject considered by the investigator, for any reason, to be an unsuitable candidate
* Female subject who is pregnant or breast-feeding or considering becoming pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Redden, MD, PhD, Study Director — Abbott
Locations (11):
- China (11):
  - Site Reference ID/Investigator# 6259, Hefei, AN
  - Site Reference ID/Investigator# 6266, Beijing
  - Site Reference ID/Investigator# 6241, Beijing
  - Site Reference ID/Investigator# 6243, Guangzhou
  - Site Reference ID/Investigator# 6247, Guangzhou
  - Site Reference ID/Investigator# 6262, Harbin
  - Site Reference ID/Investigator# 6248, Hepingjiebeikou
  - Site Reference ID/Investigator# 6250, Shanghai
  - Site Reference ID/Investigator# 6828, Shanghai
  - Site Reference ID/Investigator# 6333, Shanghai
  - Site Reference ID/Investigator# 6264, Xi'an

REFERENCES:
- [Derived] Burmester GR, Landewe R, Genovese MC, Friedman AW, Pfeifer ND, Varothai NA, Lacerda AP. Adalimumab long-term safety: infections, vaccination response and pregnancy outcomes in patients with rheumatoid arthritis. Ann Rheum Dis. 2017 Feb;76(2):414-417. doi: 10.1136/annrheumdis-2016-209322. Epub 2016 Jun 23. PMID 27338778

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo administered subcutaneously (SC) every other week (eow) for 12 weeks, followed by adalimumab 40 mg SC eow for 12 weeks.
- Adalimumab 40 mg: Adalimumab 40 mg administered subcutaneously (SC) every other week (eow) for 24 weeks.
- Adalimumab 80 mg: Adalimumab 80 mg administered subcutaneously (SC) every other week (eow) for 12 weeks, followed by adalimumab 40 mg SC eow for 12 weeks.
Period: DB Wk 0 Through 12 (Primary D/C Reasons)
Arm/Group | Placebo | Adalimumab 40 mg | Adalimumab 80 mg
Started | 60 | 121 | 121
Completed | 59 | 119 | 116
Not Completed | 1 | 2 | 5
Not completed — Adverse Event | 1 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Various | 0 | 0 | 0
Period: OL Wk 24 to End (Primary D/C Reasons)
Arm/Group | Placebo | Adalimumab 40 mg | Adalimumab 80 mg
Started | 59 | 119 | 116
Completed | 23 | 55 | 52
Not Completed | 36 | 64 | 64
Not completed — Adverse Event | 2 | 10 | 11
Not completed — Withdrawal by Subject | 15 | 19 | 25
Not completed — Lost to Follow-up | 1 | 10 | 6
Not completed — Various | 18 | 25 | 22

BASELINE CHARACTERISTICS:
Groups:
- Adalimumab 40 mg: Adalimumab 40 mg administered subcutaneously (SC) every other week (eow) for 104 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Adalimumab 40 mg | Adalimumab 80 mg | Total
Number analyzed (Participants) | 60 | 121 | 121 | 302
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 58 | 115 | 111 | 284
  >=65 years | 2 | 6 | 10 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 104 | 101 | 254
  Male | 11 | 17 | 20 | 48
Region of Enrollment [Number; unit: participants]
  China | 60 | 121 | 121 | 302

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With American College of Rheumatology (ACR)20 at Week 12 of the Double-Blind Period
Description: American College of Rheumatology (ACR) criteria improvement consisting of 20% (ACR20) reduction in tender or swollen joint counts and 20% improvement in 3 of the following 5 criteria: 1) physician's global assessment of disease activity, 2) subject's assessment of disease activity, 3) subject's assessment of pain, 4) subject's assessment of functional disability via a health assessment questionnaire, and 5) C-reactive protein at each visit. Week 12 = end of Double-Blind period.
Time Frame: Week 12
Population: Intent-to-treat population (ITT): all randomized subjects who received at least 1 dose of study drug during the double-blind portion of the study.
Measure: Number; unit: Participants
Arm/Group | Placebo | Adalimumab 40 mg | Adalimumab 80 mg
Number analyzed (Participants) | 60 | 121 | 121
Participants | 21 | 69 | 62
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 80 mg; A sample size of 42 subjects in the placebo group and 84 subjects in each of the adalimumab groups was needed to achieve 98% power to detect that the ACR20 response rate in the 80 mg adalimumab group was different from placebo and to achieve 84% power to detect that the 40 mg adalimumab group was different from placebo; Test type: Superiority or Other; p = 0.026, Cochran-Mantel-Haenszel — Each comparison was tested at the 2-sided alpha level of 0.05. Subjects with missing data were imputed to be non-responders. The overall type I error rate was preserved by a hierarchical stepwise closed testing procedure; Odds Ratio (OR) = 2.19, 95% CI [1.09 to 4.39]
Statistical Analysis 2: Comparison: Placebo vs Adalimumab 40 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.68, 95% CI [1.35 to 5.30]

2. Secondary Outcome: Number of Participants Achieving American College of Rheumatology (ACR)50/70 at Week 12 of the Double-Blind Period
Description: American College of Rheumatology (ACR) criteria improvement consisting of 50% or 70% (ACR50/70) reduction in tender or swollen joint counts and 50% or 70% improvement in 3 of the following 5 criteria: 1) physician's global assessment of disease activity, 2) subject's assessment of disease activity, 3) subject's assessment of pain, 4) subject's assessment of functional disability via a health assessment questionnaire, and 5) C-reactive protein at each visit. Week 12 = end of Double-blind period.
Time Frame: Week 12
Population: Intent-to-Treat (ITT) population (all randomized subjects who received at least 1 dose of study drug during the double-blind portion of the study), non-responder imputation (NRI; missing ACR responses imputed as non-responders).
Measure: Number; unit: Participants
Arm/Group | Placebo | Adalimumab 40 mg | Adalimumab 80 mg
Number analyzed (Participants) | 60 | 121 | 121
Participants
  ACR50 | 9 | 39 | 29
  ACR70 | 2 | 19 | 11
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40 mg; Test type: Superiority or Other; p = 0.009, Cochran-Mantel-Haenszel — The between-treatment comparison between each adalimumab group vs. placebo was performed at the 2-sided alpha = 0.05 significance level, without using a stepwise testing procedure or alpha adjustment; Percentage ACR responders at Week 12 were compared between adalimumab and placebo groups, where missing ACR responses were imputed as non-responder
Statistical Analysis 2: Comparison: Placebo vs Adalimumab 80 mg; Test type: Superiority or Other; p = 0.121, Cochran-Mantel-Haenszel

3. Secondary Outcome: Number of Participants Achieving American College of Rheumatology (ACR)20 Response Through Week 92 of Open-Label Period
Description: American College of Rheumatology (ACR) criteria improvement in a subject's disease condition versus Baseline consisting of 20% (ACR20) reduction in tender or swollen joint counts and 20/50/70% improvement in 3 of the following 5 criteria: 1) physician's global assessment of disease activity, 2) subject's assessment of disease activity, 3) subject's assessment of pain, 4) subject's assessment of functional disability via a health assessment questionnaire, and 5) C-reactive protein at each visit.
Time Frame: Week 0, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 92
Population: Intent-to-Treat (ITT) population (all randomized subjects who received at least 1 dose of study drug during the Open-Label period. Participant numbers are reduced from the Double-Blind period as not all enrolled participants in the DB period also enrolled in the OL period.
Measure: Number; unit: Participants
Groups:
- All Open-Label Adalimumab: All treatment groups participating in the Double-Blind period of the study.
Arm/Group | All Open-Label Adalimumab
Number analyzed (Participants) | 294
Participants
  Week 0 Responders (n = 293) | 152
  Week 4 Responders (n = 289) | 179
  Week 8 Responders (n = 283) | 183
  Week 12 Responders (n = 279) | 207
  Week 24 Responders (n = 208) | 153
  Week 36 Responders (n = 200) | 158
  Week 48 Responders (n = 183) | 147
  Week 60 Responders (n = 166) | 131
  Week 72 Responders (n = 150) | 108
  Week 84 Responders (n = 137) | 111
  Week 92 Responders (n = 130) | 105

4. Secondary Outcome: Number of Participants Achieving American College of Rheumatology (ACR)50 Response Through Week 92 of Open-Label Period
Description: American College of Rheumatology (ACR) criteria improvement in a subject's disease condition versus Baseline consisting of 50% (ACR50) reduction in tender or swollen joint counts and 20/50/70% improvement in 3 of the following 5 criteria: 1) physician's global assessment of disease activity, 2) subject's assessment of disease activity, 3) subject's assessment of pain, 4) subject's assessment of functional disability via a health assessment questionnaire, and 5) C-reactive protein at each visit.
Time Frame: Week 0, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 92
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | All Open-Label Adalimumab
Number analyzed (Participants) | 294
Participants
  Week 0 Responders (n = 293) | 77
  Week 4 Responders (n = 289) | 95
  Week 8 Responders (n = 283) | 103
  Week 12 Responders (n = 279) | 119
  Week 24 Responders (n = 208) | 96
  Week 36 Responders (n = 200) | 102
  Week 48 Responders (n = 183) | 94
  Week 60 Responders (n = 166) | 74
  Week 72 Responders (n = 150) | 79
  Week 84 Responders (n = 137) | 74
  Week 92 Responders (n = 130) | 69

5. Secondary Outcome: Number of Participants Achieving American College of Rheumatology (ACR)70 Response Through Week 92 of Open-Label Period
Description: American College of Rheumatology (ACR) criteria improvement in a subject's disease condition versus Baseline consisting of 70% (ACR70) reduction in tender or swollen joint counts and 20/50/70% improvement in 3 of the following 5 criteria: 1) physician's global assessment of disease activity, 2) subject's assessment of disease activity, 3) subject's assessment of pain, 4) subject's assessment of functional disability via a health assessment questionnaire, and 5) C-reactive protein at each visit.
Time Frame: Week 0, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 92
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | All Open-Label Adalimumab
Number analyzed (Participants) | 294
Participants
  Week 0 Responders (n = 293) | 32
  Week 4 Responders (n = 289) | 39
  Week 8 Responders (n = 283) | 49
  Week 12 Responders (n = 279) | 52
  Week 24 Responders (n = 208) | 39
  Week 36 Responders (n = 200) | 48
  Week 48 Responders (n = 183) | 40
  Week 60 Responders (n = 166) | 37
  Week 72 Responders (n = 150) | 30
  Week 84 Responders (n = 137) | 38
  Week 92 Responders (n = 130) | 34

6. Secondary Outcome: Mean Change in Tender Joint Count (TJC) and Swollen Joint Count (SJC) at Week 12 of the Double-Blind Period
Description: Sixty-eight or 66 joints or regions (34 or 32 per body side [hip joints excluded]) were assessed by pressure and joint manipulation on physical examination for tender joint count (TJC) or swollen joint count (SJC), respectively. Both joint tenderness and swelling were classified as either present ("1"), absent ("0"), replaced ("9"), or no assessment ("NA"). The Total TJC or SJC was derived as the sum of all 1s evaluated; the range for TJC and SJC were 0 - 68 and 0 - 66, respectively. The higher the joint count, the worse the rheumatoid arthritis. Week 12 = end of Double-Blind period.
Time Frame: Baseline, Week 12
Population: Intent-to-Treat (ITT) population (all randomized subjects who received at least 1 dose of study drug during the double-blind portion of the study), Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Placebo | Adalimumab 40 mg | Adalimumab 80 mg
Number analyzed (Participants) | 60 | 120 | 120
Joints
  TJC Week 12 | -7.0 (12.1) | -12.2 (14.9) | -8.8 (12.6)
  SJC Week 12 | -4.7 (8.7) | -8.6 (8.6) | -6.4 (6.6)

7. Secondary Outcome: Mean Change in Tender Joint Count (TJC) Through Week 92 of the Open-Label Period
Description: as for outcome 6
Time Frame: Baseline, Week 0, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 92
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | All Open-Label Adalimumab
Number analyzed (Participants) | 294
Joints
  Baseline | 22.8 (16.07)
  Week 0 (n = 293) | -9.9 (13.44)
  Week 4 (n = 289) | -12.3 (13.08)
  Week 8 (n = 283) | -13.4 (13.68)
  Week 12 (n = 279) | -14.4 (14.15)
  Week 24 (n = 208) | -16.4 (13.54)
  Week 36 (n = 200) | -16.5 (13.57)
  Week 48 (n = 183) | -17.6 (14.24)
  Week 60 (n = 166) | -17.0 (13.99)
  Week 72 (n = 150) | -18.0 (14.15)
  Week 84 (n = 137) | -18.5 (15.18)
  Week 92 (n = 130) | -18.0 (14.23)

8. Secondary Outcome: Mean Change in Swollen Joint Count (SJC) Through Week 92 of the Open-Label Period
Description: as for outcome 6
Time Frame: Baseline, Week 0, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 92
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | All Open-Label Adalimumab
Number analyzed (Participants) | 294
Joints
  Baseline | 11.2 (7.74)
  Week 0 (n = 293) | -6.9 (8.03)
  Week 4 (n = 289) | -7.4 (8.87)
  Week 8 (n = 283) | -8.3 (8.16)
  Week 12 (n = 279) | -8.8 (7.87)
  Week 24 (n = 208) | -9.3 (8.62)
  Week 36 (n = 200) | -9.3 (8.41)
  Week 48 (n = 183) | -9.7 (8.45)
  Week 60 (n = 166) | -9.0 (7.95)
  Week 72 (n = 150) | -9.2 (7.90)
  Week 84 (n = 137) | -9.5 (7.99)
  Week 92 (n = 130) | -9.5 (8.00)

9. Secondary Outcome: Mean Change in Visual Analog Scale (VAS) Score at Week 12 of the Double-Blind Period
Description: Visual analog scale (VAS) was used for the physician's (PhGA) and patient's (PGA) global assessment of disease activity and the patient's assessment of pain. PhGA assessed the patient's current status, PGA assessed status within the last 24 h, and patient's assessment of pain assessed pain status during the last week. All 3 assessments were scored on a 100 mm horizontal scale. The scores range from 0 (no symptoms) to 100 (maximum symptoms); therefore lower VAS scores represent a better disease state. Week 12 = end of Double-Blind period.
Time Frame: Baseline, Week 12
Population: Intent-to-Treat (ITT) population (all subjects who received at least 1 dose of study drug during the double-blind period), Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | Adalimumab 40 mg | Adalimumab 80 mg
Number analyzed (Participants) | 60 | 120 | 120
mm
  PhGA, Week 12 | -20.6 (19.1) | -25.1 (22.7) | -20.9 (19.7)
  Pain, Week 12 | -14.9 (26) | -22.7 (25.2) | -16.4 (22.4)
  PGA, Week 12 | -13.8 (26.2) | -23.6 (25.2) | -16.3 (25.5)

10. Secondary Outcome: Mean Change in Physician's Global Assessment of Disease Activity (Visual Analog Scale [VAS]) Through Week 92 of the Open-Label Period
Description: Visual analog scale (VAS) was used for the physician's (PhGA) and patient's (PGA) global assessment of disease activity and the patient's assessment of pain. PhGA assessed the patient's current status, PGA assessed status within the last 24 h, and patient's assessment of pain assessed pain status during the last week. All 3 assessments were scored on a 100 mm horizontal scale. The scores range from 0 (no symptoms) to 100 (maximum symptoms); therefore lower VAS scores represent a better disease state.
Time Frame: Baseline, Week 0, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 92
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | All Open-Label Adalimumab
Number analyzed (Participants) | 294
mm
  Baseline | 60.1 (16.40)
  Week 0 (n = 293) | -22.8 (20.67)
  Week 4 (n = 289) | -25.5 (21.27)
  Week 8 (n = 283) | -28.3 (22.17)
  Week 12 (n = 279) | -31.3 (21.15)
  Week 24 (n = 208) | -30.7 (20.88)
  Week 36 (n = 200) | -33.6 (21.03)
  Week 48 (n = 183) | -33.5 (20.58)
  Week 60 (n = 166) | -32.6 (21.86)
  Week 72 (n = 150) | -32.6 (22.26)
  Week 84 (n = 137) | -33.8 (20.99)
  Week 92 (n = 130) | -35.0 (19.02)

11. Secondary Outcome: Mean Change in Patient's Assessment of Pain (Visual Analog Scale [VAS]) Through Week 92 of the Open-Label Period
Description: as for outcome 10
Time Frame: Baseline, Week 0, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 92
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | All Open-Label Adalimumab
Number analyzed (Participants) | 294
mm
  Baseline | 60.5 (19.19)
  Week 0 (n = 293) | -18.7 (23.96)
  Week 4 (n = 289) | -21.1 (24.55)
  Week 8 (n = 283) | -23.3 (26.25)
  Week 12 (n = 279) | -27.1 (24.34)
  Week 24 (n = 208) | -25.4 (23.46)
  Week 36 (n = 200) | -27.4 (24.86)
  Week 48 (n = 183) | -27.0 (25.81)
  Week 60 (n = 166) | -28.0 (26.54)
  Week 72 (n = 150) | -26.4 (28.14)
  Week 84 (n = 137) | -27.8 (24.71)
  Week 92 (n = 130) | -27.1 (25.41)

12. Secondary Outcome: Mean Change in Patient's Global Assessment of Disease Activity (Visual Analog Scale [VAS]) Through Week 92 of the Open-Label Period
Description: as for outcome 10
Time Frame: Baseline, Week 0, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 92
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | All Open-Label Adalimumab
Number analyzed (Participants) | 294
mm
  Baseline | 60.7 (19.61)
  Week 0 (n = 293) | -19.0 (25.18)
  Week 4 (n = 289) | -21.0 (26.19)
  Week 8 (n = 283) | -23.6 (26.88)
  Week 12 (n = 279) | -26.3 (25.79)
  Week 24 (n = 208) | -26.6 (25.13)
  Week 36 (n = 200) | -29.8 (25.32)
  Week 48 (n = 183) | -30.5 (26.02)
  Week 60 (n = 166) | -28.7 (28.38)
  Week 72 (n = 150) | -28.7 (25.98)
  Week 84 (n = 137) | -30.5 (25.62)
  Week 92 (n = 130) | -29.6 (25.04)

13. Secondary Outcome: Mean Change in the Disability Index of the Health Assessment Questionnaire (HAQ) Scores From Baseline to Week 12 of the Double-Blind Period
Description: HAQ is a self-reported, subject-oriented outcome measure. The Standard Disability Index of HAQ for a subject is calculated as the mean of the following 8 category scores (range: 0-3): dressing and grooming, rising, eating, walking, hygiene, reach, grip, and activities. The score of each category is calculated as the maximum of the scores for the questions of that category. The Disability Index cannot be computed if the patient does not have scores for at least 6 categories. A decrease in the Disability Index = improvement in disease (0 = no difficulties). Week 12 = end of Double-Blind period.
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Adalimumab 40 mg | Adalimumab 80 mg
Number analyzed (Participants) | 60 | 120 | 120
score on a scale | -0.3 (0.7) | -0.5 (0.5) | -0.4 (0.6)

14. Secondary Outcome: Mean Change in the Disability Index of the Health Assessment Questionnaire (HAQ) Through Week 92 of the Open-Label Period
Description: HAQ is a self-reported, subject-oriented outcome measure. The Standard Disability Index of HAQ for a subject is calculated as the mean of the following 8 category scores (range: 0-3): dressing and grooming, rising, eating, walking, hygiene, reach, grip, and activities. The score of each category is calculated as the maximum of the scores for the questions of that category. The Disability Index cannot be computed if the patient does not have scores for at least 6 categories. A decrease in the Disability Index indicates an improvement in disease (0 = no difficulties).
Time Frame: Baseline, Week 0, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 92
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Open-Label Adalimumab
Number analyzed (Participants) | 294
score on a scale
  Baseline | 1.38 (0.692)
  Week 0 (n = 293) | -0.42 (0.575)
  Week 4 (n = 289) | -0.51 (0.584)
  Week 8 (n = 283) | -0.55 (0.621)
  Week 12 (n = 279) | -0.61 (0.620)
  Week 24 (n = 208) | -0.56 (0.617)
  Week 36 (n = 200) | -0.58 (0.609)
  Week 48 (n = 183) | -0.60 (0.622)
  Week 60 (n = 166) | -0.65 (0.631)
  Week 72 (n = 150) | -0.65 (0.603)
  Week 84 (n = 137) | -0.63 (0.590)
  Week 92 (n = 130) | -0.62 (0.591)

15. Secondary Outcome: Mean Change in the SF-36 Health Survey Index Physical Component Summary (PCS) and Mental Component Summary (MCS) at Week 12 of the Double-Blind Period
Description: SF-36 (v.2) is a standardized health survey consisting of 36 questions to measure functional health status. The SF-36 score has two components: physical (PCS) and mental (MCS). Summary scores are calculated using the following 8 scales: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The score for a component is an average of the individual question scores, which are scaled 0 (not functioning) to 100 (highest functioning). An increase in SF-36 PCS or MCS indicates improved health status.
Time Frame: Baseline, Week 12
Population: Intent-to-Treat (ITT) population (all randomized subjects who received at least 1 dose of study drug during the Double-Blind portion of the study), Observed cases included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Adalimumab 40 mg | Adalimumab 80 mg
Number analyzed (Participants) | 59 | 119 | 119
score on a scale
  Physical Component Score, Week 12 | 4.2 (7.1) | 5.7 (7.3) | 4.5 (7.6)
  Mental Component Score, Week 12 | 3.5 (11.8) | 4.9 (10.7) | 2.5 (12.1)

16. Secondary Outcome: Mean Change in the SF-36 Health Survey Index Physical Component Summary (PCS) Through Week 92 of the Open-Label Period
Description: as for outcome 15
Time Frame: Baseline, Week 0, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 92
Population: Intent-to-Treat (ITT) population (all randomized subjects who received at least 1 dose of study drug during the Open-Label period). Participant numbers are reduced from the Double-Blind period as not all enrolled participants in the DB period also enrolled in the OL period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Open-Label Adalimumab
Number analyzed (Participants) | 294
score on a scale
  Baseline | 32.14 (7.759)
  Week 0 (n = 293) | 5.01 (7.356)
  Week 12 (n = 283) | 7.15 (8.225)
  Week 24 (n = 208) | 6.8 (7.251)
  Week 36 (n = 200) | 7.96 (7.478)
  Week 48 (n = 183) | 8.17 (8.046)
  Week 60 (n = 166) | 8.29 (7.666)
  Week 72 (n = 150) | 7.77 (8.806)
  Week 84 (n = 137) | 8.38 (8.182)
  Week 92 (n = 130) | 8.49 (8.195)

17. Secondary Outcome: Mean Change in the SF-36 Health Survey Index Mental Component Summary (MCS) Through Week 92 of the Open-Label Period
Description: as for outcome 15
Time Frame: Baseline, Week 0, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 92
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Open-Label Adalimumab
Number analyzed (Participants) | 294
score on a scale
  Baseline | 36.50 (10.894)
  Week 0 (n = 293) | 3.74 (11.494)
  Week 12 (n = 283) | 5.73 (12.686)
  Week 24 (n = 208) | 5.22 (11.699)
  Week 36 (n = 200) | 5.51 (11.268)
  Week 48 (n = 183) | 5.29 (11.285)
  Week 60 (n = 166) | 5.56 (10.716)
  Week 72 (n = 150) | 4.75 (10.825)
  Week 84 (n = 137) | 5.09 (11.998)
  Week 92 (n = 130) | 4.14 (11.867)

ADVERSE EVENTS:
Time Frame: The duration for adverse event reporting was 92 weeks. Data from the Double-Blind period (Week 0 through Week 12) and from any adalimumab exposure (Week 0 through Week 92) were reported.
Description: AEs were recorded from the first day of Adalimumab (ADA) treatment through 70 days after the last dose of ADA. **A placebo participant during the DB period was not included in this group, as this participant discontinued from the study prior to the OL period, thus having no ADA exposure (AEs were recorded for 301 out of 302 enrolled subjects).**
Groups:
- DB Phase - Placebo EOW: Placebo administered subcutaneously every other week during Double-Blind treatment.
- DB Phase - Adalimumab 40 mg EOW: Adalimumab 40 mg administered subcutaneously every other week during Double-Blind treatment.
- DB Phase - Adalimumab 80 mg EOW: Adalimumab 80 mg administered subcutaneously every other week during Double-Blind treatment.
- Any Adalimumab: Any adalimumab exposure during the entire study, whether from Double-Blind or Open-Label treatment.
Arm/Group | DB Phase - Placebo EOW | DB Phase - Adalimumab 40 mg EOW | DB Phase - Adalimumab 80 mg EOW | Any Adalimumab
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/121 | 3/121 | 23/301
Other Adverse Events (participants affected / at risk) | 11/60 | 30/121 | 27/121 | 84/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Phase - Placebo EOW (N=60) | DB Phase - Adalimumab 40 mg EOW (N=121) | DB Phase - Adalimumab 80 mg EOW (N=121) | Any Adalimumab (N=301)
Cerebral hemorrhage (Nervous system disorders) | 0 | 0 | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Splenic lesion (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 2
Thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Disseminated tuberculosis (Infections and infestations) | 0 | 0 | 0 | 2
Lymph node tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1
Peritoneal tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 5
Tuberculoma of central nervous system (Infections and infestations) | 0 | 0 | 0 | 1
Tuberculous pleurisy (Infections and infestations) | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pulmonary hilar enlargement (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Abortion induced (Surgical and medical procedures) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Phase - Placebo EOW (N=60) | DB Phase - Adalimumab 40 mg EOW (N=121) | DB Phase - Adalimumab 80 mg EOW (N=121) | Any Adalimumab (N=301)
Injection site pruritus (General disorders) | 0 | 7 | 5 | 0
Nasopharyngitis (Infections and infestations) | 4 | 7 | 9 | 32
Upper respiratory tract infection (Infections and infestations) | 7 | 17 | 15 | 60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.